CLINICAL TRIAL: NCT04430998
Title: Efficacy of a Zinc-L-Carnosine -Based Mouth Rinse on Periodontal Tissues and Pain After Scaling and Root Planing - a Randomized Clinical Trial; a Randomized Controlled Trial
Brief Title: Efficacy of Zinc L-Carnosine Mouth Rinse
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Collaborators: Azienda Farmaceutica Italiana SRL (Industry)
Responsible Party: Principal Investigator, Chiara Occhipinti, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COCMFFP-M-01-2020
Record Dates: First submitted 2020-06-06; First posted 2020-06-16 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Periodontal Index; Pain
Keywords: Periodontal index; Pain
MeSH Terms: conditions — Pain | interventions — polaprezinc; Chlorhexidine; chlorhexidine gluconate; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zinc L-Carnosine mouth rinse (Experimental): Using undiluted 10 ml of Zinc L-Carnosine mouth rinse, retain for 60 seconds, 3 times daily
  Interventions: Drug: Zinc L-Carnosine
- Chlorhexidine (Active Comparator): Using undiluted 10 ml of Chlorhexidine mouth rinse, retain for 60 seconds, 3 times daily
  Interventions: Drug: Chlorhexidine
- Water (Placebo Comparator): Mouth rinsing with 10 ml of water, retain for 60 seconds, 3 times daily
  Interventions: Other: Water

INTERVENTIONS:
Drug: Zinc L-Carnosine — Undiluted 10 ml of Zinc L-Carnosine mouth rinse, retain for 3 minutes, 3 times daily
  Other Names: Hepilor
  Arms: Zinc L-Carnosine mouth rinse
Drug: Chlorhexidine — Undiluted 10 ml of Chlorhexidine mouth rinse, retain for 3 minutes, 3 times daily
  Other Names: Curasept
  Arms: Chlorhexidine
Other: Water — Rinse mouth with 10 ml of water, retain for 3 minutes, 3 times daily
  Arms: Water

SUMMARY:
A clinical trial to assess the effect of a Zinc-L-Carnosine-based mouth rinse on periodontal tissues and pain after scaling and root planing

DETAILED DESCRIPTION:
A randomized, double blind, 3 group parallel study with random allocation of 75 patients to any of three groups; Zinc-L-Carnosine-based mouth rinse, Chlorhexidine mouth rinse and placebo (water) control. Three days after professional oral hygiene, which aimed at the normalization of the periodontal index, the primary (HI, VAS) and secondary (mSBI; FMPS; VMI; SI) outcomes of the study are measured to obtain baseline information, and then scaling and root planing are carried out.

The participants will be advised to follow their regular oral hygiene procedures (tooth brushing) in addition to the allocated mouth rinse. They will be examined again for primary and secondary outcomes at 7 and 21 days.

Clinical evaluation:

Clinical examination of each participant will be done by a single examiner using the previously described VAS scale and a UNC periodontal probe (No. 5 explorer Hu-Friedy, Chicago, Ill). In addition to these indices, each subject will be asked to report any adverse events they have encountered during the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PSR score greater than 2 that undergo a session of scaling and root planing

Exclusion Criteria:

* Use of mouth rinses or local or general medication in the preceding three weeks
* Any condition related with allergy or sensitivity with the mouth rinses ingredients
* Systemic and chronic diseases in progress

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-06-22 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Healing Index (H.I.) | 0, 7, 21 days
  The Laundry-Turnbull and Howley index will be used to evaluate healing, considering the changes made by Pippi et al. In 2015. In particular, seven parameters will be assessed, to each of which a value of 1 or 0 will be assigned. The sum of the values will indicate the degree of healing to be compared between the different groups.
  These seven parameters are: redness of mucosa, granulation tissue, suppuration, swelling, re-epithelialization, bleeding, pain on palpation.
  Higher score means worse outcome.
Change in the Visual Analogue Scale (VAS) of pain | 0, 7, 21 days
  Participants will be asked to mark the perceived degree of pain on a scale of 100 dashes, with the lowest score being "no pain" and the highest "the worst pain".
  Higher score means worse outcome.

SECONDARY OUTCOMES:
Change in Modified Sulcus Bleeding index (Mombelli) (mSBI) | 0, 7, 21 days
  The clinical examination of each participant will be carried out by a single examiner using the UNC periodontal probe and the explorer n. 5 (Hu-Friedy, Chicago, III) to assess sulcus bleeding and assign a score: 0 absence of bleeding;
  1. presence of bleeding on probing without redness and edema;
  2. presence of bleeding on probing with redness and edema;
  3. spontaneous bleeding.
  6 sites (3 buccal + 3 lingual / palatal) are considered for each tooth.
  Higher score means worse outcome.
Change in Full Mouth Plaque Score (O'Leary) (FMPS) | 0, 7, 21 days
  Quantitative plaque index, indicates presence of plaque on teeth. Six sites (3 buccal + 3 lingual / palatal) are considered for each tooth, to which a score is given:
  0: absence of plaque
  1. one third (1/3) of the surface shows plaque
  2. two thirds (2/3) of the surface show plaque
  3. more than 2/3 of the surface shows plaque
  Higher score means worse outcome.
Change in Calculus index (Volpe-Manhold index) (VMI) | 0, 7, 21 days
  Assessment of tartar on lingual surface of lower anterior teeth, expressed in millimeters. Three measurements are taken for each tooth; mesio-lingual, central lingual and disto-lingual.
  Total score is the sum of all measurements of all six lower anterior teeth.
  Higher score means worse outcome.
Change in Stain index (Macpherson stain index) (S.I.) | 0, 7, 21 days
  Assessment of tooth staining. Expressed via score and plus signs:
  0-1 mild stains + 1.1 - 2 moderate stains ++ 2.1 - 3 heavy stains +++
  Average stain value = sum of stain scores / total number of teeth
  Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Occhipinti, Professor, Principal Investigator — University of Milan
Locations (1):
- UOC Maxillofacial Surgery and Odontology, University of Milan, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doi H, Fujiwara M, Suzuki H, Niwa Y, Nakayama M, Shikata T, Odawara S, Takada Y, Kimura T, Kamikonya N, Hirota S. Polaprezinc reduces the severity of radiation-induced mucositis in head and neck cancer patients. Mol Clin Oncol. 2015 Mar;3(2):381-386. doi: 10.3892/mco.2014.479. Epub 2014 Dec 19. PMID 25798271
- [Background] Loe H. Oral hygiene in the prevention of caries and periodontal disease. Int Dent J. 2000 Jun;50(3):129-39. doi: 10.1111/j.1875-595x.2000.tb00553.x. PMID 10967765
- [Background] Tartaglia GM, Kumar S, Fornari CD, Corti E, Connelly ST. Mouthwashes in the 21st century: a narrative review about active molecules and effectiveness on the periodontal outcomes. Expert Opin Drug Deliv. 2017 Aug;14(8):973-982. doi: 10.1080/17425247.2017.1260118. Epub 2016 Nov 20. PMID 27835926
- [Background] Van der Weijden FA, Van der Sluijs E, Ciancio SG, Slot DE. Can Chemical Mouthwash Agents Achieve Plaque/Gingivitis Control? Dent Clin North Am. 2015 Oct;59(4):799-829. doi: 10.1016/j.cden.2015.06.002. PMID 26427569
- [Background] Omatsu T, Naito Y, Handa O, Mizushima K, Hayashi N, Qin Y, Harusato A, Hirata I, Kishimoto E, Okada H, Uchiyama K, Ishikawa T, Takagi T, Yagi N, Kokura S, Ichikawa H, Yoshikawa T. Reactive oxygen species-quenching and anti-apoptotic effect of polaprezinc on indomethacin-induced small intestinal epithelial cell injury. J Gastroenterol. 2010 Jul;45(7):692-702. doi: 10.1007/s00535-010-0213-9. Epub 2010 Feb 20. PMID 20174833